CLINICAL TRIAL: NCT03309397
Title: Stress Urinary Incontinence in Teenage Girls Practicing Sports
Brief Title: Stress Urinary Incontinence of Sporting Teenager
Acronym: INCREASE
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: INCREASE ( 29BRC17.0114)
Record Dates: First submitted 2017-10-06; First posted 2017-10-13 (Actual); Last update posted 2019-08-12 (Actual); Status verified 2019-08

CONDITIONS: Urinary Incontinence, Stress
Keywords: adolescent sports
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Physical activity and sport are beneficial to the cardiovascular system, the musculoskeletal system and many chronic pathologies. The High Authority of Health (HAS) recommends a regular practice. However, depending on the discipline and level of practice, it may be responsible for traumatic injuries, degenerative musculoskeletal injuries, overtraining, eating disorders or cardiovascular events. It also promotes urinary stress incontinence, by increasing intra-abdominal pressure in some situations.

The prevalence of urinary leakage in the athlete depends of the practiced physical activity. A classification of the sports activities can be carried out according to the risk of increased pressures on the pelvic floor:

* high-risk sports: trampoline (10.17), acrobatic gymnastics, aerobics, athletics (jumping hedges, heights, triple jump), horse riding, basketball, volleyball, handball, martial arts;
* moderate-risk sports: tennis, skiing ...
* low risk sports: walking, swimming, cycling, rollerblading, golf ... In sports, urinary incontinence also depends of the practiced movements (jumps, abdominal exercises ...), and the occurence of sports activity. This disorder has even become one of the concerns of federal sports authority (INSEP).

However, there is no data regarding stress incontinence of sports teenagers found n the literature on

ELIGIBILITY:
Inclusion Criteria:

* Between 10 and 18 years
* Consultation in medical sporting center

Exclusion Criteria:

* urge incontinence

Ages: 10 Years to 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Sporting Young Girl
Sampling Method: Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2018-01-17 (Actual); Primary Completion 2019-01-16 (Actual); Study Completion 2019-01-16 (Actual)

PRIMARY OUTCOMES:
prevalence of stress urinary incontinence in adolescent girls engaged in extra-scholar sports | Day 0
  answer by YES or NO to the question

SECONDARY OUTCOMES:
Delay of urinary incontinence according to the first menstruations | 12 months
  answer to question about the delay of first menstruations on day: less than 6 months- between 6 and 12 months- more than 12 months.

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest, Brest, France